CLINICAL TRIAL: NCT03287011
Title: Efficacy of Shoplaq® Disclosing Toothpaste in Removing Dental Plaque: A Randomized Controlled Clinical Trial.
Brief Title: Efficacy of a Plaque Disclosing Toothpaste on Home Oral Hygiene Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Segi University (Other)
Responsible Party: Principal Investigator, Avita Rath, Dr, Segi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SUKD
Record Dates: First submitted 2017-09-11; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Chronic Gingivitis, Plaque Induced
Keywords: dental plaque; tooth pastes; oral hygiene
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: interventional preventive trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Toothpaste tubes will be masked so the care provider would not know which tube he/she allocating to the participants as well the outcome assessor would be masked from both groups ( test and control) so data is assessed unbiased.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control tooth paste (Active Comparator): controlled fluoridated toothpaste will be provided for brushing to both the groups initially
  Interventions: Other: Colgate toothpaste
- Shoplaque tooth paste (Experimental): Fluoridated toothpaste with organic plaque disclosing dye will be given to the test group second visit
  Interventions: Other: Shoplaq toothpaste

INTERVENTIONS:
Other: Shoplaq toothpaste — ACTIVE INGREDIENT Sodium Monofluorophosphate 1000 PPM INGREDIENTS Precipitated Calcium Carbonate, Sorbitol, Glycerin, Precipitated Silica, Sodium Carboxy Methyl Cellulose, Sodium Benzoate, DM Water, Colour CI-45410, Holy Basil Oil, Neem Oil, Citrus Oil, Thymol Oi, Clove Oil, Piper Betel Leaf Oil, Tea Tree Oil, Eucalyptus Oil, Peppermint Oil, Spearmint Oil.
  Dye containing tooth paste for disclosing plaque and efficient brushing for better oral health.
  Arms: Shoplaque tooth paste
Other: Colgate toothpaste — fluoridated
  Arms: Control tooth paste

SUMMARY:
Plaque accumulation on tooth and gingival surfaces is a causative factor for oral diseases such as demineralization, dental caries, gingivitis, and periodontitis.

Tooth brushing and flossing have been the cornerstone of oral hygiene and health. However, the high incidence and prevalence of gum problems in both the developed and developing world show these mechanical routines are not enough. Furthermore, many patients find it difficult to comply with this daily regime of brushing and flossing. Consistent with problems associated with maintaining oral health, periodontal disease is one of the most common chronic infections in adults. According to Philstrom, et al. up to 90% of the world's population has or will suffer from periodontal disease.Thus, the maintenance of an adequate level of plaque control by the individual through his or her daily oral hygiene is vital to prevent and control periodontal disease. Studies demonstrate that poor oral hygiene is widespread with about 60% of plaque found on the surfaces of the teeth after brushing. This may be due to the lack of manipulative skills, lack of motivation and compliance.Hence, increasing education and improving brushing technique by improving oral hygiene products is one way to enhance plaque removal in everyday brushing. The ability to see plaque while brushing will enhance patient's awareness and encourage them to be more thorough when performing oral hygiene.

DETAILED DESCRIPTION:
Plaque accumulation on tooth and gingival surfaces is a causative factor for oral diseases such as demineralization, dental caries, gingivitis, and periodontitis. 1 Thus, the maintenance of an adequate level of plaque control by the individual through his or her daily oral hygiene is vital to prevent and control periodontal disease which can result in tooth mobility and tooth loss. 2 Tooth brushing and flossing have been the cornerstone of oral hygiene and health.2 However, the high incidence and prevalence of gum problems in both the developed and developing countries show these mechanical routines are not enough. 1 Studies demonstrate that poor oral hygiene is widespread with about 60% of plaque found on the surfaces of the teeth after brushing.3 Furthermore, many patients find it difficult to comply with this daily regimen of brushing and flossing. 2 This may be due to the lack of manipulative skills, lack of motivation and compliance. 2 According to an overview of the challenges in dental public health in Malaysia by Allan Kah, he stated that only 26% of 15-19-year-old and only 5% of 35-44-year-olds have been reported to have healthy periodontal tissues. 4 Studies such as the one done by Deliargyris, showed that periodontal disease was associated with the enhanced systemic inflammatory response with various mediators. Thus, it may contribute to systemic diseases. For example, periodontal disease has been linked to atherosclerosis via an increased level of serum C-reactive protein, a marker for inflammation and a high-risk factor for coronary artery disease.5 Hence, there is a need to increase education and improve brushing technique. This can be done by improving oral hygiene products by incorporating a plaque disclosing dye in the toothpaste.1 The ability to see plaque while brushing will enhance patient's awareness and encourage them to be more thorough when performing oral hygiene. 1 Previous studies done by the Department of Orthodontics, University of Illinois have shown that using a toothpaste with a plaque indicating dye such as PlaqueHD® to disclose plaque while brushing resulted in more than four times as much plaque elimination between visits (51.3% reduction, p = 0.015) than participants using only the placebo toothpaste (8.3% reduction, p=0.189). 1 However, one of the limitations of the product used in that study is the high cost of the toothpaste and the difficulty in obtaining the toothpaste in South East Asia.Hence, the present study aims to assess the efficacy of a plaque disclosing toothpaste that is easily available and affordable which was developed with the Health Promotion Board of Singapore, named Shoplaq® in reducing dental plaque.

ELIGIBILITY:
Inclusion Criteria:

* Students of SEGi must be aged 18 to 25 years with chronic generalized gingivitis 2)
* With no known systemic illness.
* Minimum of 12 anterior teeth present (canine to canine) in both upper and lower arches

Exclusion Criteria:

* Participants who are pregnant or nursing.
* A dental student or faculty or dental staff member.
* Who have been on antibiotics within two weeks prior to examination.
* Having dry mouth syndrome or significant food allergies.
* Have undergone any dental procedures or oral prophylaxis within 30 days prior to testing

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Plaque removal efficacy of a disclosing toothpaste | from Baseline to 1 year
  Silness and Loe plaque index
Assessment of prevalence and severity of gingivitis in individuals who use the disclosing toothpaste | from Baseline to 1 year
  Loe and Silness gingival index

SECONDARY OUTCOMES:
digital image analysis | from Baseline to 1 year
  MATLAB software for digital image analysis
adverse effects | baseline to 1 year
  To record any side effects or adverse effects of the toothpaste seen by the patient or
  clinician. soft tissue changes, taste alteration
patient perceived outcomes | baseline to 1 year
  self-administered questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Avita Rath, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
article with study description and result
Supporting Information: Study Protocol, CSR
Time Frame: July 2018
Access Criteria: through journal publication